CLINICAL TRIAL: NCT06753669
Title: Mothers' Action Project for Child Health
Acronym: MAP-CH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Alison Karasz, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00000666; UH3DE030070 (NIH)
Record Dates: First submitted 2024-10-27; First posted 2024-12-31 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Dental Caries; Obesity Risk
Keywords: early childhood caries; child obesity; social network intervention
MeSH Terms: conditions — Dental Caries; Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Referrals to vetted dentists, educational materials on child feeding and oral health, in person health education sessions and social network building
  Interventions: Behavioral: health education and social network building
- Control Arm (Placebo Comparator): The control arm will receive referrals to vetted dentists and educational materials on child feeding and oral health.
  Interventions: Behavioral: dental referral and educational materials

INTERVENTIONS:
Behavioral: health education and social network building — The investigators will use techniques from the social network literature to build each treatment group as a cohesive social network and will diffuse educational messages through these groups. Educational materials and vetted dentist referrals, plus navigation to dentist visits, will be provided.
  Arms: Intervention arm
Behavioral: dental referral and educational materials — Control arm will receive a referral to vetted dentist and educational materials on child health
  Arms: Control Arm

SUMMARY:
This randomized controlled trial will recruit Bangladeshi mothers and their young children into a 12 month intervention that provides child health and oral health education and seeks to build social networks among mothers.

DETAILED DESCRIPTION:
MAP-CH is a cluster randomized clinical trial. A total of 66 proximally dwelling clusters of approximately 7 mothers will be randomized 1:1 to the intervention and control arms (33 clusters/arm). One child per family will be enrolled, resulting in a total sample size of 460. The target population of this study is low-income SA mothers of young children aged 12-66 months.

Recruitment: To identify eligible families for recruitment, the MAP-CH research staff will conduct a Mapping Project. Outreach workers will identify clusters of eligible families living close together in SA neighborhoods. Accompanied by local contacts project staff will visit homes of potential participants and assess eligibility and recruit eligible consenting mothers.

Intervention: Mothers assigned to the intervention group will participate in a 12-month, multi-session, group-based intervention. Intervention meetings will take place in participant homes and will be led in Bengali (or the language spoken by that cluster), by a skilled bilingual facilitator from our research staff. The intervention is designed to: 1) improve knowledge, attitudes, and behaviors related to reducing dietary sugar; and 2) increase maternal assertiveness and parenting skills related to healthy feeding; and 3) build lasting social networks supportive of these norms and behaviors among participants. Eighteen sessions will be delivered over 12 months.

Control group: Mothers assigned to the control arm will receive a series of packages and mailings.

Data collection: Interviews will be conducted in the home, by RAs at T1/Baseline, T2 (12months' post baseline) and T3 (18 months' post baseline). Data collected at each interview includes anthropometric data collection; and questionnaires/interviews. Social network data will also be collected at T1, 3M, 6M, T1, and T3. Dental caries assessments will occur at baseline and T3.

Analyses: The primary outcome is reduced d2-4mfs increment at 18 months' post baseline in the intervention compared to the control group. A secondary outcome is reduced weight gain velocity. Other outcomes include servings of sweetened foods and beverages, servings of junk food, use of bottles, maternal feeding behaviors, oral hygiene, and dental utilization. The investigators will also evaluate potential mediators and moderators of treatment impact including knowledge, assertiveness, depression, household empowerment, and social network quality.

ELIGIBILITY:
Inclusion Criteria:

* Mother:

  * Age >=18;
  * Speaks and reads/writes Bengali or Hindi/Urdu;
  * Mother born in a South Asian country;
  * Mother is primary caretaker of child
* Child:

  * Aged >=12 and <=48 months
  * Has Medicaid or CHIP (NYS health plan for low income families not qualifying for Medicaid)

Exclusion Criteria:

* Mother:

  * Unable to provide informed consent,
  * Lack of availability--either plans to travel for > 1 month during 12 month initial study period or other barriers to attendance;
  * Mother has exclusionary health condition--either intellectual/cognitive or medical.
* Child:

  * Weighed < 5lbs at birth,
  * Has an exclusionary health condition and/or is taking long term (>1 m) antibiotics;
  * Not the youngest eligible child in family

Ages: 12 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 460 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
NIDCR ECC Collaborative Criteria Dental Exam | 18 months
  The investigators will assess 18 month incidence in dental caries using dental hygienist exams at baseline and 18 months post baseline. The exams will be conducted in the home, in the knee to knee position or on the floor, using artificial light and a front plane mirror. The teeth will be dry brushed and wiped. An explorer will be used to remove debris to visualize the tooth surface except as specified for the assessment of hardness. No magnification will be allowed. The examiner will use a trained recorder.

SECONDARY OUTCOMES:
Weight Gain Velocity | 18 months
  We will measure child weight and height/length at 0, 12 and 18 months. Research staff will obtain weight and height data at baseline, 12 and 18 m. For children under 24 months of age, two supine measures will be taken using infantometers (Seca 417), to the nearest 0.1 cm. For children ≥24 months, a stadiometer will be used. If measurements differ by +/- 0.5 cm., a third measure will be taken, and the means averaged. Research quality scales will be used to assess weight. Primary outcome is change in weight/height over 18 months.
Infant Feeding Styles Questionnaire--Adapted | 18 months
  This measure assesses maternal feeding style, including pressured feeding. The original measure has been heavily adapted for the current population. The scale includes 19 items. The score ranges from 0 to 76 with a higher score indicating more problematic feeding styles.
Oral Hygiene and Dental Utilization Questionnaire | 18 months
  This 25 Item inventory, adapted for a previous study with a similar population, includes subscales covering the following domains: holding a bottle, sleeping with a bottle, tooth brushing, toothpaste, tap water, dental visits.
Food frequency Questionnaire | 18 months
  This seven day food frequency questionnaire has been adapted for use in the current study. It includes a variety of subscales focusing on food items relevant to weight gain and dental health including breast milk, formula, cows milk, sweetened beverages, sweets, junk food/snacks, and fruits/vegetables.
Dental utilization | 18 months
  Presence or absence of a dental visit AND # dental visits between baseline and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Alison Karasz, Principal Investigator — UMass Chan

IPD SHARING:
Plan to Share IPD: Yes
Demographics, social network, and outcome data
Supporting Information: SAP
Time Frame: Data will be available indefinitely as soon as all study analyses are complete
Access Criteria: Qualified researcher with a clear analysis plan